CLINICAL TRIAL: NCT04901663
Title: Comparison of Vonoprazan and Amoxicillin Dual Therapy With Standard Triple Therapy With Proton Pump Inhibitor for Helicobacter Pylori Eradication; a Randomized Control Trial
Brief Title: Vonoprazan in Helicobacter Pylori Treatment an RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Bader Faiyaz Zuberi, Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAD-VPZ-001
Record Dates: First submitted 2021-05-18; First posted 2021-05-25 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Helicobacter Pylori Infection
Keywords: helicobacter pylori; Vonoprazan; potassium-competitive acid inhibitor
MeSH Terms: interventions — Omeprazole; Capsules; Clarithromycin; Amoxicillin

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omeprazole Group (Active Comparator): Omeprazole 20 mg BD Amoxicillin 1000 mg BD Clarithromycin 500 mg BD
  Interventions: Drug: Omeprazole 20 MG Capsule; Amoxicillin 1000 MG; Clarithromycin 500 MG
- Vonoprazan Group (Experimental): Vonoprazan 20 mg BD Amoxicillin 1000 mg BD
  Interventions: Drug: Vonoprazan 20 MG; Amoxicillin 1000 MG

INTERVENTIONS:
Drug: Omeprazole 20 MG Capsule; Amoxicillin 1000 MG; Clarithromycin 500 MG — Orally twice daily for 2 weeks
  Other Names: Omeprazole Group
  Arms: Omeprazole Group
Drug: Vonoprazan 20 MG; Amoxicillin 1000 MG — Orally twice daily for 2 weeks
  Other Names: Vonoprazan Group
  Arms: Vonoprazan Group

SUMMARY:
RCT for comparison of Standard Triple therapy (Omeprazole+Amoxil+Clarithromycin) for H Pylori erradication with Vonoprazan+Amoxil dual therapy.

DETAILED DESCRIPTION:
OBJECTIVE To compare the efficacy of Vonoprazan based dual treatment versus PPI based treatment for the eradication of Helicobacter pylori infection.

OPERATIONAL DEFINITION

Helicobacter Pylori infection: Hp infection will be labelled by any one of following investigation:

* Helicobacter Pylori Stool Antigen
* Histopathology on Giemsa Stain

MATERIAL AND METHODS:

Study Design: Randomized control trial. Setting: This study will be conducted in the Medical OPD and Medical Unit 1 of Dr. Ruth K.M. Pfau, Civil Hospital Karachi affiliated with Dow University of Health Sciences

DATA COLLECTION PROCEDURE:

All patients presenting to the OPD or Medical Unit 1 of Dr. Ruth KM Pfau, Civil Hospital Karachi and fulfilling the inclusion criteria will be included after taking informed consent.

The participants will be randomly allocated to 2 groups with help of random number table and will be treated for 2 weeks.

Group A: will be given:

Capsule Amoxicillin 1 gm twice daily Tablet Clarithromycin 500 mg twice a day Capsule Omeprazole 20 mg twice a day

Group B will be given:

Capsule Amoxicillin 1 gm twice daily Tablet Vonoprazan 20 mg twice a day Confirmation of Hp eradication will be done by stool Hp antigen test 4 weeks after completion of treatment.

DATA ANALYSIS Data will be stratified according to age & gender. Frequency of gender & mean (SD) of age will be compared between groups using Pearson's Chi-square test and Student's t-test respectively. Frequency of Hp eradication between two groups will be compared using Pearson's chi-square test. A p value < .05 will be taken as significant.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter Pylori Positive by any one of following:

Histopathology by Giemsa Stain Stool Antigen

Exclusion Criteria:

* • Previous surgery of the stomach such as partial gastrectomy.

  * Allergy to any of the antibiotics used in the study.
  * Intake of antibiotics, PPIs, corticosteroids, or nonsteroidal anti-inflammatory drugs within the last 2 weeks.
  * Pregnant or lactating females.
  * Alcohol abuse or drug addiction.
  * Severe neurological or psychiatric disorder.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2021-08-13 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Helicobacter Pylori Eradication | 4 weeks
  Stool Heliobacter Pylori Antigen = Negative

CONTACTS AND LOCATIONS:
Overall Officials: Bader F Zuberi, FCPS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dr Ruth KM Pfau Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abadi ATB, Ierardi E. Vonoprazan and Helicobacter pylori Treatment: A Lesson From Japan or a Limited Geographic Phenomenon? Front Pharmacol. 2019 Apr 5;10:316. doi: 10.3389/fphar.2019.00316. eCollection 2019. PMID 31024299
- [Result] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631
- [Result] Burucoa C, Axon A. Epidemiology of Helicobacter pylori infection. Helicobacter. 2017 Sep;22 Suppl 1. doi: 10.1111/hel.12403. PMID 28891138
- [Result] Crowe SE. Helicobacter pylori Infection. N Engl J Med. 2019 Mar 21;380(12):1158-1165. doi: 10.1056/NEJMcp1710945. No abstract available. PMID 30893536
- [Result] Munoz N, Sanchez-Delgado J, Baylina M, Lopez-Gongora S, Calvet X. Prevalence of Helicobacter pylori resistance after failure of first-line therapy. A systematic review. Gastroenterol Hepatol. 2018 Dec;41(10):654-662. doi: 10.1016/j.gastrohep.2018.06.014. Epub 2018 Sep 1. English, Spanish. PMID 30180998
- [Result] Ke H, Li J, Lu B, Yang C, Wang J, Wang Z, Liu L, Chen Y. The appropriate cutoff gastric pH value for Helicobacter pylori eradication with bismuth-based quadruple therapy. Helicobacter. 2021 Feb;26(1):e12768. doi: 10.1111/hel.12768. Epub 2020 Oct 21. PMID 33089598
- [Result] Wang YC, Chen YP, Ho CY, Liu TW, Chu CH, Wang HY, Liou TC. The Impact of Gastric Juice pH on the Intraluminal Therapy for Helicobacter pylori Infection. J Clin Med. 2020 Jun 14;9(6):1852. doi: 10.3390/jcm9061852. PMID 32545856
- [Result] Murakami K, Sakurai Y, Shiino M, Funao N, Nishimura A, Asaka M. Vonoprazan, a novel potassium-competitive acid blocker, as a component of first-line and second-line triple therapy for Helicobacter pylori eradication: a phase III, randomised, double-blind study. Gut. 2016 Sep;65(9):1439-46. doi: 10.1136/gutjnl-2015-311304. Epub 2016 Mar 2. PMID 26935876
- [Result] Yamada S, Kawakami T, Nakatsugawa Y, Suzuki T, Fujii H, Tomatsuri N, Nakamura H, Sato H, Okuyama Y, Kimura H, Yoshida N. Usefulness of vonoprazan, a potassium ion-competitive acid blocker, for primary eradication of Helicobacter pylori. World J Gastrointest Pharmacol Ther. 2016 Nov 6;7(4):550-555. doi: 10.4292/wjgpt.v7.i4.550. PMID 27867688
- [Result] Suzuki H, Mori H. World trends for H. pylori eradication therapy and gastric cancer prevention strategy by H. pylori test-and-treat. J Gastroenterol. 2018 Mar;53(3):354-361. doi: 10.1007/s00535-017-1407-1. Epub 2017 Nov 14. PMID 29138921
- [Result] Kato M, Ota H, Okuda M, Kikuchi S, Satoh K, Shimoyama T, Suzuki H, Handa O, Furuta T, Mabe K, Murakami K, Sugiyama T, Uemura N, Takahashi S. Guidelines for the management of Helicobacter pylori infection in Japan: 2016 Revised Edition. Helicobacter. 2019 Aug;24(4):e12597. doi: 10.1111/hel.12597. Epub 2019 May 20. PMID 31111585